CLINICAL TRIAL: NCT04764812
Title: Determination of Risk Factors and Awareness Associated With Development of Neuromuscular Scoliosis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Halic University (Other)
Collaborators: Medipol University (Other); Istanbul Rumeli University (Other)
Responsible Party: Sponsor
Other Study IDs: HUEK96-28
Record Dates: First submitted 2021-02-18; First posted 2021-02-21 (Actual); Last update posted 2022-02-21 (Actual); Status verified 2022-02

CONDITIONS: Neuromuscular Scoliosis; Deformity
Keywords: neuromuscular diseases; cerebral palsy; awareness; risk factors
MeSH Terms: conditions — Congenital Abnormalities; Neuromuscular Diseases; Cerebral Palsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Neuromuscular diseases caused by disruption of the normal conduction relationship between nerve system, neuromuscular junction, and muscles cause scoliosis as a secondary deformity. Neuromuscular scoliosis progresses due to muscle weakness and characteristic features of disease. The risk of complications associated with increased progression. Morbidity and mortality caused by scoliosis in neuromuscular diseases can be reduced by increasing the knowledge and awareness of the caregivers and physiotherapists. In this study, it was aimed to determine the risk of neuromuscular scoliosis and the factors which can cause in children with disabilities. It is also aimed to reveal inferences related to education levels, awareness of caregivers and professionals working in this field to determine cases with a high risk of scoliosis. Thus, it is expected to leading future research to develop preventive treatment approaches. For this purpose, 288 children who are diagnosed with the neuromuscular disease between 3-18 years of age, attending Rehabilitation Center in Istanbul and willing to participate in the research permitted by their caregiver will be included in this study. Cerebral Palsy Follow-Up Program (CPUP), Parents and Professionals Awareness Questionnaire related to Neuromuscular Scoliosis which is prepared by researchers, Early Onset Scoliosis 24 Questionnaire, Scoliosis Research Society 22 Questionnaire to assess QoL, demographic and clinical data also will collect for all sample. Patients will be examined for musculoskeletal system, scoliosis analysis will be performed radiologically. Data obtained to determine the problems, risk factors, and awareness of the caregivers and physiotherapists will be analyzed statistically.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed with neuromuscular disease or cerebral palsy
* receiving treatment at a rehabilitation center in Istanbul
* willing to participate in the research and permitted by their caregiver

Exclusion Criteria:

* Spinal infections, tumors, trauma
* Trauma history of lower extremity

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: -3-18 years patients who have neuromuscular scoliosis and various skeletal deformities due to neuromuscular disease or cerebral palsy.
Sampling Method: Non-Probability Sample
Enrollment: 288 (Estimated)
Dates: Start 2021-03-01 (Actual); Primary Completion 2022-09-20 (Estimated); Study Completion 2022-09-26 (Estimated)

PRIMARY OUTCOMES:
Cerebral Palsy Follow-Up Program (CPUP) Assessment Form | baseline
  Assessment form consisted pyhsical examination of pain, spasticity, range of motion, muscle strength, gross motor funtion stage, functional mobility, postural abilitis of patients in lying and sitting position, postural quality in sitting and standing position, screening spinal or other musculoskeletal deformities, assessment of orthotics, wheelchair or other mobility assistance if there is any that patients wearing/using.
Parents and Professionals Awareness Questionnaire related to Neuromuscular Scoliosis | baseline
  Parents and professionals knowledge and approaches to the neuromuscular scoliosis, investigate their prevention strategies.The questionnaire developed by the researchers and doesn't have a scoring system meaning better or worse outcomes.
Early Onset Scoliosis 24 Questionnaire | baseline
  The EOSQ-24 represents a subjective, parent-based, and self-report questionnaire. It includes 11 separate items in 24 questions. The domains are general health, pain, pulmonary function, mobility, physical function, daily living, fatigue, emotion, parental burden, financial burden, and satisfaction. Each question rated using a 5-point Likert scale. Total score obtain by adding domains. Higher scores indicates better qualitiy of life.
Scoliosis Research Society 22 Questionnaire | baseline
  SRS-22 questionnaire was developed by SRS to evaluate health-related quality of life (HRQL) in patients with adolescent idiopathic scoliosis (AIS) and the Turkish version was validated in 2005. The SRS-22 questionnaire consists of 22 items Likert type scale that allows scoring between 1-5 for each question. SRS-22 has five domains including function, pain, mental health, self-image and satisfaction. Subgroups can be evaluated separately, or the total score is obtained by summing up the scores from all questions. The total score of each section ranges from 5 to 25, only the section evaluating satisfaction from the treatment is in the range of 2-10. Scoring is obtained by dividing the total score of each section by the number of questions in that section. Higher scores indicate better quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Özge Ökçü, MSc., Principal Investigator — Istanbul Rumeli University; Hande Tunc, MSc., Principal Investigator — Halic University; Ahsen Buyukaslan, PhD.(c), Principal Investigator — Medipol University; Hürriyet Yılmaz, Prof.Dr., Study Director — Halic University
Locations (1):
- Rehabilitation Center, Istanbul, İ̇stanbul, Turkey (Türkiye)